CLINICAL TRIAL: NCT04338204
Title: Observational Study of Tofacitinib in Ulcerative Colitis in Sweden (ODEN)
Brief Title: Observational Study To Assess The Effectiveness and Treatment Adherence Of Tofacitinib of Ulcerative Colitis In Clinical Practice In Sweden
Acronym: ODEN
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921366; ODEN (Other: Alias Study Number)
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed tofacitinib: Patients with a confirmed diagnosis of ulcerative colitis with confirmed active disease (biomarker or endoscopy) initiating tofacitinib as per the Swedish summary of product characteristics (SmPC).
  Interventions: Drug: tofacitinib

INTERVENTIONS:
Drug: tofacitinib — Observational study

SUMMARY:
This is a prospective observational study using data from an existing, ongoing National Swedish registry (SWIBREG). This study is designed to assess the effectiveness and treatment adherence of tofacitinib on clinical disease activity parameters in patients with ulcerative colitis in Swedish clinical practice. The study will also assess treatment adherence of tofacitinib using the Swedish Prescribed Drug Register.

ELIGIBILITY:
Inclusion Criteria:

* The assignment of the patient to tofacitinib is not decided in advance by the protocol but falls within clinical practice and the prescription of the medicine is done according to the SmPC and is clearly separated from the decision to include the patient in the study.
* The patient must sign the informed consent before enrollment in the study. The informed consent permits extraction of data from SWIBREG at baseline and during the duration of the study. For patients not registered in SWIBREG, they must complete all SWIBREG consents and registration at the time of treatment initiation. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Patients, male or female, must be 18 years old or above.
* The patient must have active disease as confirmed by fecal calprotectin >250 mg/kg or endoscopic assessment corresponding to a Mayo endoscopic subscore ≥2 not more than 4 weeks prior onset to the initiation of tofacitinib treatment. This inclusion criteria applies also to patients that have already been enrolled in the study.

Exclusion Criteria:

* The patient is enrolled in a clinical trial in which the treatment of ulcerative colitis is dictated by a study protocol. If the patient is participating in another ongoing observational study (non-interventional), the patient may be included in this observational study.
* Patients that fulfill any of the contraindications according to the latest version of the SmPC. Any SmPC label updates will be communicated to all study sites.
* For whatever reason the physician feels the patient unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of ulcerative colitis, ≥18years of age, with confirmed active disease (biomarker or endoscopy) initiating tofacitinib as per the Swedish summary of product characteristics (SmPC)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants in Remission as Measured by Partial Mayo Score | Week 52
  Clinical Remission is defined as a partial score of <2 points with 0 points regarding rectal bleeding.

SECONDARY OUTCOMES:
Proportion of Participants who are taking tofacitinib | Baseline, Weeks 8, 16, 52, 104
Proportion of Participants in Clinical Remission Based on Total Mayo Score | Weeks 8, 16, 52, and 104
  Clinical Remission is defined as a total Mayo score of ≤2 points with no individual subscore exceeding 1 point, with 0 points regarding rectal bleeding.
Proportion of Participants in Clinical Response Based on Total Mayo Score | Weeks 8, 16, 52, and 104
  Clinical Response is defined as a total Mayo score decrease of ≥3 points and a decrease of ≥30% from baseline, with a decrease of ≥1 point on the rectal bleeding subscore or an absolute rectal bleeding score of ≤1
Proportion of Participants in Clinical Remission Based on Partial Mayo Score | Weeks 8, 16, 52 and 104
  Clinical Remission is defined as a partial Mayo score <2 points with 0 points regarding rectal bleeding.
Proportion of Participants in Clinical Response Based on Partial Mayo Score | Weeks 8, 16, 52 and 104
  Clinical Response is defined as a partial Mayo score decrease of ≥2 points and reduction of at least 25% in partial Mayo (pMayo) score from baseline with an accompanying decrease in rectal bleeding subscore of ≥1 point or absolute rectal bleeding subscore of ≤1 point
Proportion of Participants in Steroid-Free Clinical Remission | Baseline, weeks 8, 16, 52, and 104
  Steroid-Free Clinical Remission is defined by a total Mayo Score who did not require any corticosteroid treatment during the period ≥4 weeks prior to the visit (for all patients and for those treated with corticosteroids at baseline)
Change from Baseline in Total Mayo Score | Baseline, Weeks 8, 16, 52, and 104
Change From Baseline In Partial Mayo Score | Baseline, Weeks 8, 16, 52 and 104
Change From Baseline In Level of Fecal Calprotectin (f-calprotectin) | Baseline, Weeks 8, 16, 52 and 104
  Fecal calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Higher values indicate more serious inflammation.
Proportion of Responders defined by a Fecal Calprotectin (f-calprotectin) Reduction of ≥50%, ≥75% or ≥90% | Weeks 8, 16, 52, and 104
  Fecal calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Higher values indicate more serious inflammation.
Change from Baseline of C-Reactive Protein (CRP) | Baseline, Weeks 8, 16, 52, and 104
Proportion of Participants In Sustained Remission (Partial Mayo score) | Week 8 To Weeks 16, 52 and 104
Proportion of Participants In Sustained Remission (Partial Mayo score) | Week 16 To Weeks 52 and 104
Proportion of Participants in Sustained Steroid Free Remission (Partial Mayo Score) (for all patients and for those treated with corticosteroids at baseline) | Weeks 16 through 52 and at Week 104
Proportion of Participants in Endoscopic Remission, Mucosal Healing or Endoscopic Response | Week 8, 16, 52 and 104
  Endoscopic remission is defined as a subscore of 0. Mucosal healing is defined as a subscore of 0-1. Endoscopic response is defined as a subscore reduction from baseline of ≥1.
Proportion of Participants in Sustained Endoscopic Remission, Mucosal Healing or Endoscopic Response | Week 8 to Week 16, 52 and 104
  Endoscopic remission is defined as a subscore of 0. Mucosal healing is defined as a subscore of 0-1. Endoscopic response is defined as a subscore reduction from baseline of ≥1.
Proportion of Participants in Sustained Endoscopic Remission, Mucosal Healing or Endoscopic Response | Week 16 to 52 and at Week 104
  Endoscopic remission is defined as a subscore of 0. Mucosal healing is defined as a subscore of 0-1. Endoscopic response is defined as a subscore reduction from baseline of ≥1.
Proportion of Participants in Sustained Steroid Free Remission (Partial Mayo Score) (For All Participants and for Those Treated With Corticosteroids at Baseline) and Endoscopic Remission, Mucosal Healing or Endoscopic Response | Week 16 to 52 and 104
  Endoscopic remission is defined as a subscore of 0. Mucosal healing is defined as a subscore of 0-1. Endoscopic response is defined as a subscore reduction from baseline of ≥1.
Change From Baseline In Inflammatory Bowel Disease Fatigue (IBD-F) Score | Baseline, Weeks 8, 16, 52 and 104
Change From Baseline In EuroQol 5 Dimensions 5 Levels (EQ5D-5L) | Baseline, Weeks 8, 16, 52, and 104
Change From Baseline In Short Health Scale (SHS) | Baseline, Weeks 8, 16, 52 and 104
Proportion of Participants Who Had a Colectomy | Weeks 8, 16, 52, and 104
Comparison of Response and Remission (Partial Mayo Score) Based on the Extent of Ulcerative Colitis According To the Montreal Classification | Weeks 8, 16, 52 and 104
Proportion of Participants In Sustained Remission (Total Mayo score) | Week 16 To Weeks 52 and 104
Proportion of Participants In Sustained Remission (Total Mayo score) | Week 8 To Weeks 16, 52 and 104
Proportion of Participants in Sustained Steroid Free Remission (Total Mayo Score) (For All Participants and for Those Treated With Corticosteroids at Baseline) and Endoscopic Remission, Mucosal Healing or Endoscopic Response | Week 16 to 52 and 104
  Endoscopic remission is defined as a subscore of 0. Mucosal healing is defined as a subscore of 0-1. Endoscopic response is defined as a subscore reduction from baseline of ≥1.
Proportion of Participants in Sustained Steroid Free Remission (Total Mayo Score) (for all patients and for those treated with corticosteroids at baseline) | Weeks 16 through 52 and at Week 104
Comparison of Response and Remission (Total Mayo Score) Based on the Extent of Ulcerative Colitis According To the Montreal Classification | Weeks 8, 16, 52 and 104
Proportion of Participants in Steroid-Free Clinical Remission | Baseline, weeks 8, 16, 52, and 104
  Steroid-Free Clinical Remission is defined by a partial Mayo Score who did not require any corticosteroid treatment during the period ≥4 weeks prior to the visit (for all patients and for those treated with corticosteroids at baseline)
Proportion of participants reaching f-calprotectin below 250 mg/kg of those that had f-calprotectin above 250 mg/kg at baseline | Baseline, week 8, 16, 52 and 104
  Fecal calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Higher values indicate more serious inflammation.
Portion of participants with dose change of tofacitinib | Week 8, 16, 52 and 104
Portion of participants with a termination of tofacitinib | Week 8, 16, 52 and 104
Portion of participants with dose and dose changes of tofacitinib and corticosteroids | Week 8, 16, 52 and 104
Proportion of particpants with changes in rectal bleeding and stool frequency | Baseline, Week 2
  Proportion of patients with improvement in rectal bleeding and stool frequency with a change in baseline sub score 1
Proportion of participants with changes in EQ5D and SHS | Baseline, Week 2
Proportion of particpants with rectal bleeding and stool frequency sub score indicative of mild disease | Baseline, Week 2
Proportion of participants with stool frequency and rectal bleeding subscore of 0 | Baseline, Week 2
Proportion of participants with mild abdominal pain | Baseline, week 2, 8, 16, 52 and 104
Proportion of participants with no abdominal pain | Baseline, week 2, 8, 16, 52 and 104
Proportion of participants with no bowel urgency | Baseline, Weeks 2, 8, 16, 52 and 104.
Proportion of participants with reduction of ≥ 1 point from baseline rectal bleeding and stool frequency sub score | Baseline, Week 2
Proportion of patients achieving symptomatic remission | Baseline, weeks 2, 8, 16, 52 and 104.
  Symptomatic remission is defined as a total sum of 0 of the to Mayo sub-scores stool frequency(SF) and rectal bleeding (RB)
Proportion of patients achieving symptomatic remission stratified on steroid use at baseline or not. | Baseline, weeks 2, 8, 16, 52 and 104
Proportion of patients achieving symptomatic response | Baseline, weeks 2, 8, 16, 52 and 104
  Symptomatic response is defined as a decrease of at least 50% of the sum of the Mayo-sub-scores stool frequency (SF) and rectal bleeding (RB).
Proportion of patients achieving symptomatic response stratified on steroid use at baseline | Baseline, weeks 2, 8, 16, 52 and 104
Proportion of patients in steroid-free clinical remission (pMayo and full Mayo score)stratified based on steroid use at baseline or not. | Baseline, weeks 8, 16, 52 and 104
  Steroid-Free Clinical Remission is defined by a partial Mayo Score who did not require any corticosteroid treatment during the period ≥4 weeks prior to the visit (for all patients and for those treated with corticosteroids at baseline)
Change from baseline in bowel urgency (as measured by SCCAI) | Weeks 2, 8, 16, 52 and 104
  SCCAI is the Simple Clinical Colitis Activity Index bowel urgency sub-score used to assess the bowel urgency.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Sweden (17):
  - Ulf Eriksson, Alingsås
  - Medicinkliniken, Södra Älvsborgs Sjukhus Borås, Brämhultsvägen 53, Borås
  - Gävle Hospital, Gävle
  - SU/Sahlgrenska, Gastroenterologi & Hepatologi, Gothenburg
  - Medicinkliniken, Länssjukhuset Ryhov, Sjukhusgatan, Jönköping
  - Daniel Molin, Kristianstad
  - Shiprock Consulting AB,, Lidingö
  - Mag-Tarmmedicinska kliniken, Universitetssjukhuset i Linköping, Linköping
  - Region skåne, Skånes Universitetssjukhus, Malmo
  - Medicinmottagning 4, Medicinska Kliniken, Universitetssjukhuset Örebro, Örebro
  - Stockholm Gastro Center, Stockholm
  - Ersta Sjukhus, Medicinkliniken, Fjällgatan 44, Stockholm
  - Karolinska Universitetssjukhuset i Solna, Eugeniavägen 3, B4-09,, Stockholm
  - Danderyds Hospital, Stockholm
  - Medicinkliniken, Umeås Universitetssjukhus, Umeå
  - Specialmedicin, Akademiska Sjukhuset, Sjukhusvägen ing 40, Uppsala
  - Medicinmottagningen gastroenterologi, Västmanlands sjukhus, Västerås

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Nyberg L, Halfvarson J, Soderling J, Olen O, Strid H, Hedin CRH, Jonsdottir SB, Hjortswang H, Jaghult S, Cappelleri JC, Henrohn D, Seddighzadeh M, Marsal J, Grip O; SWIBREG ODEN Study Group. Prospective observational study of tofacitinib in ulcerative colitis - analysis of clinical data, fatigue and health-related quality of life during the induction phase. Therap Adv Gastroenterol. 2025 Jun 16;18:17562848251343427. doi: 10.1177/17562848251343427. eCollection 2025. PMID 40535533
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921366